CLINICAL TRIAL: NCT01377467
Title: A Phase 3, Investigator-initiated, Randomized, Open-label Single-center Study of the Effect of Denosumab on the Prevention of Bone Mineral Density Loss After Renal Transplantation
Brief Title: Denosumab for Prevention of Osteoporosis in Renal Transplant Recipients
Acronym: POSTOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rudolf Wuethrich (Other)
Responsible Party: Sponsor-Investigator, Rudolf Wuethrich, Professor and Director, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UZH-NEP 2.1
Record Dates: First submitted 2011-06-20; First posted 2011-06-21 (Estimated); Results first posted 2016-04-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Osteoporosis; Chronic Kidney Disease
Keywords: Osteoporosis; Osteopenia; Denosumab; Transplantation; Kidney
MeSH Terms: conditions — Osteoporosis; Renal Insufficiency, Chronic; Bone Diseases, Metabolic | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab (Experimental): 60 mg denosumab s.c. at baseline and after 6 months
  Interventions: Drug: Denosumab (Prolia)
- Control (No Intervention): No treatment

INTERVENTIONS:
Drug: Denosumab (Prolia) — 60 mg s.c. injection at baseline and after 6 months
  Other Names: Prolia
  Arms: Denosumab

SUMMARY:
The primary objective of the study is to examine the effect of denosumab on lumbar spine bone mineral density (BMD) after one year of treatment in newly transplanted renal allograft recipients. Secondary endpoints include BMD changes at the total hip and the femoral neck, changes in body height, changes in bone mineral metabolism parameters, incidence of fractures, and allograft function at one year. Safety measurements include the occurrence of rejection episodes, infectious complications, graft loss and mortality.

* Trial with medicinal product

DETAILED DESCRIPTION:
Renal allograft recipients are at high risk to suffer a substantial loss of bone mineral density (BMD) within the first year after kidney transplantation. This loss of BMD correlates with an increased risk for the development of osteoporosis or worsening of pre-existing osteopenia/osteoporosis, heightening the risk for the subsequent occurrence of fractures. Renal allograft recipients are often treated with calcium and vitamin D preparations to prevent BMD loss. The addition of bisphosphonates can further improve BMD. However, bisphosphonates are potentially nephrotoxic and promote adynamic bone disease, and are therefore not regularly prescribed.

Receptor Activator of Nuclear factor- Kappa-B Ligand (RANKL) is a key molecule mediating development, activity, and survival of osteoclasts. Osteoporosis results in part from increased osteoclastic bone resorption, and therefore the inhibition of RANKL activity has become an obvious therapeutic strategy to prevent bone mineral density (BMD) loss and the development of osteoporosis.

The novel anti-osteoporotic drug denosumab (trade name Prolia®) is a fully human monoclonal antibody against RANKL. By inhibiting the development and the activity as well as reducing the survival of osteoclasts it decreases bone resorption and increases bone density.

The hypothesis of the present study is that denosumab has a beneficial effect on the loss of BMD in the first year after renal transplantation. The preservation of BMD is a surrogate parameter, generally predicting subsequent improvements in the occurrence rate of fractures. The hypothesis will be tested by studying the effect of denosumab on BMD in newly transplanted renal allograft recipients.

The purpose of the present trial is to study the effect of denosumab on BMD in kidney allograft recipients. The study participants will be treated for 1 year, receiving a total of 2 injections of the standard 60 mg dose at baseline and at 6 months.

Ninety sequential renal allograft recipients will be randomized 1:1 to receive two subcutaneous 60 mg denosumab injections within 14 days and 6 months following renal transplantation, or no treatment. All patients will also receive oral standard treatment with 1000 mg calcium plus 800 IU vitamin D.

ELIGIBILITY:
The key inclusion criteria are:

1. Male or female adult de novo kidney, kidney-pancreas or kidney-islet, or kidney-liver transplant recipients
2. Functioning graft within 28 days after transplantation (creatinine having decreased to <200 micromol/l without the need for dialysis)
3. Being on standard triple immunosuppression including a calcineurin antagonist (cyclosporine or tacrolimus), mycophenolate (MMF or MPA) and steroids, with or without induction treatment with basiliximab or anti-thymocyte globulin

Key exclusion criteria are:

1. Age <18 years
2. Rising creatinine after initial drop <200 micromol/l or creatinine >200 micromol/l at baseline
3. Evidence of early acute rejection, either suspected clinically and/or proven by biopsy
4. Presence of severe osteoporosis as evidenced by a T score <-4 at the hip, femoral neck or any of the 4 vertebrae L1 to L4
5. Evidence of severe hyper- or hypoparathyroidism (iPTH >800 ng/l or <10 ng/l)
6. Hypocalcemia (total calcium <1.8 mmol/l) or hypercalcemia (total calcium >2.7 mmol/l)
7. Steroid-free de novo immunosuppression scheme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf P Wuthrich, MD, Principal Investigator — Division of Nephrology, University Hospital, Zurich
Locations (1):
- Division of Nephrology, University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bonani M, Frey D, Brockmann J, Fehr T, Mueller TF, Saleh L, von Eckardstein A, Graf N, Wuthrich RP. Effect of Twice-Yearly Denosumab on Prevention of Bone Mineral Density Loss in De Novo Kidney Transplant Recipients: A Randomized Controlled Trial. Am J Transplant. 2016 Jun;16(6):1882-91. doi: 10.1111/ajt.13692. Epub 2016 Feb 29. PMID 26713403
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 20, 2011, to May 2, 2014. Patients were randomized after 15.7 ± 6.4 days after transplantation.
Period: Overall Study
Arm/Group | Denosumab | Control
Started | 46 | 44
Completed | 46 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized patients with a functioning graft
Groups:
- Total: Total of all reporting groups
Arm/Group | Denosumab | Control | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (16.0) | 52.9 (14.0) | 50.9 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 19 | 19 | 38
Region of Enrollment [Number; unit: participants]
  Switzerland | 46 | 44 | 90
Number of osteopenic patients [Number; unit: participants]
  Yes | 16 | 25 | 41
  No | 30 | 19 | 49
Number of osteoporotic patients [Number; unit: participants]
  Yes | 3 | 6 | 9
  No | 43 | 38 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in BMD at the Total Lumbar Spine From Baseline to Month 12
Description: The total lumbar spine BMD was measured via Dual Energy X-ray Absorptiometry (DXA) and was expressed in g/cm2 hydroxylapatite
Time Frame: Baseline and month 12
Population: The intention-to-treat (ITT) population was used for the primary efficacy analysis, i.e. all subjects were included that have been randomized to the control group or to the denosumab group. Missing values were replaced with a last-value-carried-forward approach (LVCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 4.5 (3.8) | -0.3 (5.1)
Statistical Analysis 1: Comparison: Denosumab vs Control; We calculated that a sample size of 43 patients per group would provide a statistical power of 86% to detect a 4% difference in the percentage change of areal BMD at the total lumbar spine at 12 months, using a two-sided t-test with an α-level of 0.05 and assuming a mean ± SD change of 4 ± 6% in the denosumab group and 0 ± 6% in the control group. To account for a dropout rate of 5%, it was planned to randomize a total of 90 patients; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 5.059, 95% CI 2-sided [3.137 to 6.980], Standard Error of Mean 0.967 — Percentage change in BMD was compared between the two treatment groups while controlling for the effects of baseline BMD

2. Secondary Outcome: Percent Change in BMD at the Total Hip From Baseline to Month 12
Description: The total hip BMD was measured via Dual Energy X-ray Absorptiometry (DXA) and was expressed in g/cm2 hydroxylapatite
Time Frame: Baseline and month 12
Population: The intention-to-treat (ITT) population was used for the analysis of this endpoint, i.e. all subjects were included in the analysis that have been randomized to the control group or to the denosumab group. Missing values were replaced with a last-value-carried-forward approach (LVCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 2.3 (3.7) | 0.5 (4.2)
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.035, ANCOVA; Mean Difference (Final Values) = 1.895, 95% CI 2-sided [0.132 to 3.659], Standard Error of Mean 0.887 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Change in BMD at the Femoral Neck From Baseline to Month 12
Description: The total femoral neck BMD was measured via Dual Energy X-ray Absorptiometry (DXA) and was expressed in g/cm2 hydroxylapatite
Time Frame: Baseline and month 12
Population: The intention-to-treat (ITT) was used for the analysis of this endpoint, i.e. all subjects were included in the analysis that have been randomized to the control group or to the denosumab group. Missing values were replaced with a last-value-carried-forward approach (LVCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 1.1 (4.7) | 0.8 (6.0)
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.380, ANCOVA; Mean Difference (Final Values) = 1.059, 95% CI 2-sided [-1.329 to 3.447], Standard Error of Mean 1.201 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change in BMD at the Total Lumbar Spine From Baseline to Month 6
Description: The total lumbar spine BMD was measured via DXA and was expressed in g/cm2 hydroxylapatite.
Time Frame: Baseline and month 6
Population: The intention-to-treat was used for the analysis of this endpoint, i.e. all subjects were included in the analysis that have been randomized to the control group or to the denosumab group. Missing values were replaced with a last-value-carried-forward approach (LVCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 2.9 (3.3) | -1.5 (4.1)
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 4.567, 95% CI 2-sided [2.975 to 6.178], Standard Error of Mean 0.806 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Change in BMD at the Total Hip From Baseline to Month 6
Description: The total hip BMD was measured via DXA and was expressed in g/cm2 hydroxylapatite
Time Frame: Baseline and month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 1.4 (2.4) | -0.3 (1.4)
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.009, ANCOVA; Mean Difference (Final Values) = 1.756, 95% CI 2-sided [0.440 to 3.072], Standard Error of Mean 0.662 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Change in BMD at the Femoral Neck From Baseline to Month 6
Description: The femoral neck BMD was measured via DXA and was expressed in g/cm2 hydroxylapatite
Time Frame: Baseline and month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 46 | 44
percent change | 1.0 (4.0) | -0.8 (5.4)
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.064, ANCOVA; Mean Difference (Final Values) = 2.035, 95% CI 2-sided [-0.122 to 4.193], Standard Error of Mean 1.085 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Beta-CTX at Baseline and Months 3, 6 and 12
Description: Blood concentrations of beta-CTX (microgram/L)
Time Frame: baseline, month 3, month 6, and month 12
Population: For this endpoint, an available case analysis was performed, i.e., all randomised patients with valid data at all time points were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: microgram/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 42 | 42
microgram/L
  baseline | 0.635 [0.508 to 0.741] | 0.772 [0.665 to 0.878]
  month 3 | 0.129 [0.037 to 0.221] | 0.590 [0.498 to 0.682]
  month 6 | 0.204 [0.077 to 0.330] | 0.612 [0.485 to 0.739]
  month 12 | 0.389 [0.154 to 0.623] | 0.794 [0.559 to 1.028]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p < 0.001, repeated measures GLM; between-subjects effect = 10.466 — Within-subjects effect: p=0.007. Time*treatment interaction: p=0.002. The a priori threshold for statistical significance is <0.05

8. Secondary Outcome: P1NP at Baseline and Months 3, 6 and 12
Description: Blood concentrations of P1NP were measured in microgram/L
Time Frame: baseline, month 3, month 6, and month 12
Population: For this endpoints, an available case analysis was performed, i.e., all randomised patients with valid data at all time points were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: microgram/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 42 | 41
microgram/L
  baseline | 61.222 [47.974 to 74.470] | 77.808 [64.399 to 91.217]
  month 3 | 40.976 [19.801 to 62.152] | 108.699 [87.266 to 130.13]
  month 6 | 35.347 [11.525 to 59.169] | 107.072 [82.962 to 131.18]
  month 12 | 57.953 [33.685 to 82.221] | 132.439 [107.876 to 157.0]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p < 0.001, repeated measures GLM; between-subjects effect = 275622.016 — Within-subjects effect: p<0.001. Time*treatment interaction: p=0.012. The a priori threshold for statistical significance is <0.05

9. Other Pre Specified Outcome: Blood Levels of Calcium (mmol/L) at Baseline and Months 0.5, 1, 2, 3, 6, 12
Description: Blood levels of calcium (mmol/L) were measured at baseline and at months 0.5, 1, 2, 3, 6, and 12
Time Frame: baseline, months 0.5, 1, 2, 3, 6, 12
Population: For this endpoints, an available case analysis was performed, thus all randomised patients with valid data at all time points were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 30 | 35
mmol/L
  baseline | 2.320 [2.245 to 2.395] | 2.317 [2.247 to 2.386]
  month 0.5 | 2.131 [2.049 to 2.214] | 2.405 [2.329 to 2.481]
  month 1 | 2.293 [2.231 to 2.356] | 2.444 [2.387 to 2.502]
  month 2 | 2.420 [2.355 to 2.485] | 2.480 [2.419 to 2.540]
  month 3 | 2.404 [2.327 to 2.481] | 2.461 [2.390 to 2.532]
  month 6 | 2.463 [2.404 to 2.522] | 2.453 [2.399 to 2.508]
  month 12 | 2.480 [2.421 to 2.538] | 2.509 [2.455 to 2.563]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.014, repeated measures GLM; between-subjects effect = 0.717 — Within-subjects effect: p<0.001. Time*treatment interaction: p<0.001. The a priori threshold for statistical significance is <0.05

10. Other Pre Specified Outcome: Blood Levels of Phosphate (mmol/L) at Baseline and Months 0.5, 1, 2, 3, 6, 12
Description: Blood levels of phosphate (mmol/L) were measured at baseline and at months 0.5, 1, 2, 3, 6, 12
Time Frame: baseline, months 0.5, 1, 2, 3, 6, 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 32 | 36
mmol/L
  baseline | 0.582 [0.506 to 0.657] | 0.586 [0.514 to 0.657]
  month 0.5 | 0.525 [0.436 to 0.613] | 0.714 [0.631 to 0.798]
  month 1 | 0.605 [0.519 to 0.691] | 0.726 [0.645 to 0.807]
  month 2 | 0.726 [0.659 to 0.793] | 0.812 [0.749 to 0.875]
  month 3 | 0.742 [0.673 to 0.812] | 0.776 [0.711 to 0.842]
  month 6 | 0.804 [0.727 to 0.880] | 0.849 [0.777 to 0.921]
  month 12 | 0.842 [0.737 to 0.948] | 0.902 [0.802 to 1.002]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.068, repeated measures GLM; between-subjects effect = 0.707 — Within-subjects effect: p<0.001. Time*treatment interaction: p=0.047. The a priori threshold for statistical significance is <0.05

11. Other Pre Specified Outcome: Blood Levels of PTH (ng/L) at Baseline and Months 3, 6, and 12
Description: Blood levels of PTH (ng/L) were measured at baseline and at months 3, 6, and 12
Time Frame: baseline and months 3, 6, and 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 40 | 40
ng/L
  baseline | 163.110 [115.906 to 210.314] | 147.300 [100.096 to 194.504]
  month 3 | 173.573 [130.141 to 217.004] | 111.563 [68.131 to 154.994]
  month 6 | 157.043 [117.092 to 196.993] | 99.420 [59.469 to 139.371]
  month 12 | 106.650 [85.078 to 128.222] | 100.705 [79.133 to 122.277]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.114, repeated measures GLM; between-subjects effect = 99952.126 — [estimate comment as in outcome 10, analysis 1]

12. Other Pre Specified Outcome: 25-OH-vitamin D3
Description: Blood levels of 25-OH-vitamin D3 were measured as microgramm/L
Time Frame: baseline, months 3, 6, and 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: microgramm/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 41 | 40
microgramm/L
  baseline | 17.378 [14.690 to 20.067] | 18.058 [15.336 to 20.779]
  month 3 | 21.632 [19.604 to 23.659] | 22.903 [20.850 to 24.955]
  month 6 | 24.395 [21.418 to 27.373] | 26.728 [23.713 to 29.742]
  month 12 | 28.546 [25.890 to 31.202] | 28.358 [25.669 to 31.046]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.578, repeated measures GLM; between-subjects effect = 84.830 — Within-subjects effect: p<0.001. Time*treatment interaction: p=0.593. The a priori threshold for statistical significance is <0.05

13. Other Pre Specified Outcome: 1,25-(OH)2 Vitamin D3
Description: Blood levels of 1,25-(OH)2 vitamin D3 were measured as ng/L
Time Frame: baseline, months 3, 6, and 12
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/L
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 36 | 34
ng/L
  baseline | 29.556 [21.977 to 37.134] | 34.171 [26.373 to 41.969]
  month 3 | 60.533 [52.678 to 68.389] | 55.276 [47.193 to 63.360]
  month 6 | 54.175 [46.883 to 61.467] | 58.074 [50.570 to 65.577]
  month 12 | 47.208 [39.902 to 54.515] | 51.494 [43.976 to 59.013]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.607, repeated measures GLM; between-subjects effect = 248.686 — Within-subjects effect: p<0.001. Time*treatment interaction: p=0.296. The a priori threshold for statistical significance is <0.05

14. Other Pre Specified Outcome: Percent Change From Baseline in Total Volumetric Bone Mineral Densitiy (Tot.vBMD) at the Distal Tibia
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal tibia and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 2.2 [0.7 to 3.2] | -0.3 [-3.3 to 2.7]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.019, Wilcoxon (Mann-Whitney); z value = -2.342

15. Other Pre Specified Outcome: Percent Change From Baseline in Cortical Volumetric Bone Mineral Densitiy (Ct.vBMD) at the Distal Tibia
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal tibia and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 0.1 [-0.5 to 1.4] | -0.5 [-2.0 to 0.1]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.042, Wilcoxon (Mann-Whitney); z value = -2.049

16. Other Pre Specified Outcome: Percent Change From Baseline in Trabecular Volumetric Bone Mineral Densitiy (Tb.vBMD) at the Distal Tibia
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal tibia and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 1.8 [1.3 to 4.2] | 1.1 [-2.5 to 4.1]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.371, Wilcoxon (Mann-Whitney); z value = -0.937

17. Other Pre Specified Outcome: Percent Change From Baseline in Cortical Thickness (Ct.Th) at the Distal Tibia
Description: Cortical thickness was measured via HR-pQCT (Xtreme CT) at the distal tibia and was expressed as mm.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 2.8 [1.4 to 8.0] | -0.9 [-5.9 to 1.6]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney); z value = -2.752

18. Other Pre Specified Outcome: Percent Change From Baseline in Total Volumetric Bone Mineral Densitiy (Tot.vBMD) at the Distal Radius
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal radius and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 1.3 [-1.9 to 2.2] | -1.6 [-5.2 to 0.7]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.031, Wilcoxon (Mann-Whitney); z value = -2.166

19. Other Pre Specified Outcome: Percent Change From Baseline in Cortical Volumetric Bone Mineral Densitiy (Ct.vBMD) at the Distal Radius
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal radius and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | -0.1 [-1.8 to 1.3] | -0.9 [-2.7 to 0.4]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.212, Wilcoxon (Mann-Whitney); z value = -1.288

20. Other Pre Specified Outcome: Percent Change From Baseline in Trabecular Volumetric Bone Mineral Densitiy (Tb.vBMD) at the Distal Radius
Description: Volumetric BMD (vBMD) was measured via HR-pQCT (Xtreme CT) at the distal radius and was expressed as mg HA/cm3.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 2.4 [1.1 to 4.1] | 0.2 [-9.4 to 3.1]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.108, Wilcoxon (Mann-Whitney); z value = -1.640

21. Other Pre Specified Outcome: Percent Change From Baseline in Cortical Thickness (Ct.Th) at the Distal Radius
Description: Cortical thickness was measured via HR-pQCT (Xtreme CT) at the distal radius and was expressed as mm.
Time Frame: Baseline and month 12
Population: Subgroup of patients (n=24) who participated in the HR-pQCT (Xtreme CT) subprotocol.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab | Control
Number analyzed (Participants) | 10 | 14
Percent change | 0.9 [-6.0 to 2.0] | -3.6 [-7.7 to -1.3]
Statistical Analysis 1: Comparison: Denosumab vs Control; Test type: Superiority or Other; p = 0.048, Wilcoxon (Mann-Whitney); z value = -1.991

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Denosumab | Control
Serious Adverse Events (participants affected / at risk) | 31/46 | 29/44
Other Adverse Events (participants affected / at risk) | 45/46 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denosumab (N=46) | Control (N=44)
Urinary tract infection (Infections and infestations) | 11 (12) | 2 (6)
Transplant pyelonephritis (Infections and infestations) | 3 (3) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
CMV viremia (Infections and infestations) | 1 (1) | 5 (5)
Flu-like disease (Infections and infestations) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lymphocele (Blood and lymphatic system disorders) | 6 (6) | 6 (7)
Acute rejection (Immune system disorders) | 2 (2) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Diabetes (post-transplant) (Endocrine disorders) | 0 (0) | 1 (1)
Surgical intervention (Surgical and medical procedures) | 0 (0) | 2 (2)
Functional decline of transplant function (Renal and urinary disorders) | 4 (5) | 1 (1)
Transplant ureter stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Peripheral arterial vascular disease (Vascular disorders) | 0 (0) | 1 (1)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Transplant artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterus myomatosus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Retinitis (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence (Surgical and medical procedures) | 0 (0) | 1 (1)
Bilateral nephrectomy of polycystic kidneys (Renal and urinary disorders) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 3 (3) | 0 (0)
Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 1 (1) | 0 (0)
Neck/back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized weakness (General disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Ureteral leakage (Renal and urinary disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 3 (3) | 0 (0)
Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Choledocholithiasis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyponatremia (Endocrine disorders) | 1 (1) | 0 (0)
Infection without focus (Infections and infestations) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transplant reflux testing (Surgical and medical procedures) | 1 (1) | 0 (0)
Selective ureteral sampling (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Urethral stricture (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Denosumab (N=46) | Control (N=44)
Urinary tract infections (Infections and infestations) | 12 (39) | 5 (19) — Cystitis (bladder infection)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 4 (4)
Hypocalcemia (Endocrine disorders) | 12 (12) | 1 (1) — Transient, asymptomatic hypocalcemia defined as total serum calcium <1.9 mmol/L
Thrombosis (Vascular disorders) | 1 (1) | 4 (4)
Aphtous stomatitis (Infections and infestations) | 2 (3) | 3 (3)
Fever (General disorders) | 1 (1) | 3 (4)
Hemorrhoids (Gastrointestinal disorders) | 2 (3) | 4 (4)
Sore throat (Infections and infestations) | 4 (4) | 5 (5)
Tremor (Nervous system disorders) | 2 (2) | 7 (7)
Exanthema (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (4)
Headache (General disorders) | 4 (4) | 3 (3)
Muscle pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Neck/back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 3 (3)
Rhinorrhea (General disorders) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 3 (6) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Alopecia (General disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (7) | 2 (2)
Fecal blood (Gastrointestinal disorders) | 3 (3) | 0 (0)
Edema (General disorders) | 5 (6) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (5) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes